CLINICAL TRIAL: NCT06549322
Title: The Efficacy of Exercise Timing - Effects of Resistance Exercise on Eating Behavior and Energy Metabolism
Brief Title: Timing and Resistance Exercise: Impact on Eating and Metabolism
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Normal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 202401HM008
Record Dates: First submitted 2024-08-08; First posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Circadian Rhythm; Energy Balance; Appetitive Behavior; Food Reward
Keywords: resistance exercise; energy expenditure
MeSH Terms: conditions — Appetitive Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The exercise in morning (Experimental): Resistance exercises are in the following order: squat, bench press, deadlift. Each exercise consists of 3 sets with 7 repetitions, using a load of 70% 1RM with 60 sec of rest between sets.
  Interventions: Other: The exercise in morning
- The exercise in evening (Experimental): Resistance exercises are in the following order: squat, bench press, deadlift. Each exercise consists of 3 sets with 7 repetitions, using a load of 70% 1RM with 60 sec of rest between sets.
  Interventions: Other: The exercise in evening
- The control in all day (No Intervention): Sit and rest in the morning and evening during the day.

INTERVENTIONS:
Other: The exercise in morning — Resistance exercises are in the following order: squat, bench press, deadlift. Each exercise consists of 3 sets with 7 repetitions, using a load of 70% 1RM with 60 sec of rest between sets.
  Exercise timing: AM 11:00-11:30
  Arms: The exercise in morning
Other: The exercise in evening — Resistance exercises are in the following order: squat, bench press, deadlift. Each exercise consists of 3 sets with 7 repetitions, using a load of 70% 1RM with 60 sec of rest between sets.
  Exercise timing: PM 05:00-05:30
  Arms: The exercise in evening

SUMMARY:
Exercise timing (morning or evening) for optimal weight control is a research topic urgently addressed by scholars in the relevant field. Due to the better control of energy metabolism and physical activity levels in the morning, existing research on resistance exercise and eating behavior primarily focuses on experiments conducted in the morning, with only one study in the afternoon. No research has yet compared the potential differences between morning and evening resistance exercise. A one-year study aims to investigate the impact of morning and evening resistance exercise on physiological metabolism and eating behavior. Eighteen healthy male participants will be randomly assigned to a crossover design study, including AM exercise, PM exercise, and control (rest condition) trials. Variables including subjective appetite, appetite hormones (ghrelin, peptide YY), food preferences, ad libitum eating, dietary records, energy expenditure, and PBMCs circadian rhythm genes will be measured. This preliminary study through a multidimensional observation, the results will contribute to understanding the potential differences and mechanisms of morning and evening resistance exercise on physiological metabolism and eating behavior. In practical applications, conducting resistance exercise in the evening or at night aligns better with current lifestyles. The findings of this study can support the optimization of exercise benefits by validating the choice of exercise timing.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-30
* weight stable for at least 6 months

Exclusion Criteria:

* Obesity (BMI > 30 kg/m² or body fat percentage > 25%)
* Hypertension (blood pressure over 140/90 mmHg)
* Heart disease
* Cancer
* Liver or kidney diseases
* Any other conditions that could potentially influence the study's outcomes

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Subjective appetite Subjective appetite Subjective appetite Subjective appetite Subjective appetite Subjective appetite | 3 hours during each study intervention
  The appetite perceptions are obtained through a 0-100 mm visual analog scale. The variables assessed include perceptions of hunger (i.e., "How hungry do you feel?"), satisfaction (i.e., "How satisfied do you feel?"), fullness (i.e., "How full do you feel?"), prospective food consumption (i.e., "How much do you think you can eat?"), and nausea (i.e., "How nauseous do you feel?"), with 0 indicating "not at all" and 100 signifying "extremely.".
Change in acyl-Ghrelin | 3 hours during each study intervention
  acyl-Ghrelin in pg/mL
Change in PYY | 3 hours during each study intervention
  PYY in pg/mL
Change in Leptin | 3 hours during each study intervention
  Leptin in pg/mL
Change in lactate | 3 hours during each study intervention
  lactate in mmol/L
Change in PBMCs circadian rhythm genes | 3 hours during each study intervention
  Circadian rhythm genes in PBMC will be measured, such as Bmal1, Clock, Per1, Per2, Per3, Cry1, Cry2, Cry3, and Tbp in arbitrary units.
Energy intake | The Before day, the durning day, and the day following the experiment.
  Participants will be required to record their diet for the day before, the current day, and the day following the experiment.
  The energy intake include absolute energy intake and relative energy intake .
Energy expenditure | The Before day, the durning day, and the day following the experiment.
  Participants will record energy expenditure during resistance exercise, with non-exercise energy expenditure measured using an accelerometer.

SECONDARY OUTCOMES:
Explicit liking | 3 hours during each study intervention
  A visual analog scale ranging from 0 to 100 mm is utilized to evaluate the question, "How pleasant would it be to taste some of this food now?" with 0 indicating "not at all" and 100 signifying "extremely."
Explicit wanting | 3 hours during each study intervention
  A visual analog scale ranging from 0 to 100 mm is utilized to evaluate the question, "How much do you want some of this food now?" with 0 indicating "not at all" and 100 signifying "extremely."
Implicit wanting | 3 hours during each study intervention
  Participants are given a set of food image pairs and are asked to select their preference by answering the question, "Which food do you desire the most at the moment?". The implicit wanting calculation involves further consideration of response time data based on preference choices using a standardized equation.
Relative preference | 3 hours during each study intervention
  Participants are given a set of food image pairs and are asked to select their preference by answering the question, "Which food do you desire the most at the moment?". The relative preference is the sum of the times each type of food is chosen, with a maximum value of 48 and a minimum value of 0.
Taste appeal bias | 3 hours during each study intervention
  Taste preference (savoury or sweet) is calculated by subtracting the mean savory scores from the mean sweet scores. Positive values suggest a preference for sweet foods, while negative scores indicate a preference for savory foods, and a score of 0 signifies an equal preference between taste categories.
Fat appeal bias | 3 hours during each study intervention
  Fat preference (high or low) is calculated by subtracting the mean low-fat scores from the mean high-fat scores. Positive values suggest a preference for high-fat foods, while negative scores indicate a preference for low-fat or savory foods, and a score of 0 signifies an equal preference between fat content.
change in Cortisol | 3 hours during each study intervention
  Cortisol mcg/dL
change in complete blood count | 3 hours during each study intervention
  change in complete blood count cells/L
change in growth hormone | 3 hours during each study intervention
  growth hormone pmol/L

CONTACTS AND LOCATIONS:
Overall Officials: Hung-wen Liu, Ph.D., Principal Investigator — National Taiwan Normal University
Locations (1):
- National Taiwan Normal University, Taipei, Taiwan